CLINICAL TRIAL: NCT00874198
Title: European Multicenter Study on the Prediction of Outcome in Patients With Idiopathic Normal Pressure Hydrocephalus
Brief Title: European Study on Prediction of Outcome in Patients With Idiopathic Normal Pressure Hydrocephalus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: International Neuroscience Institute Hannover (Other)
Collaborators: Sahlgrenska University Hospital (Other); Department of Neurology and Neurosurgery,Westeinde Hospital, Den Haag (Unknown); Uppsala University Hospital (Other); University of Copenhagen (Other); Unfallkrankenhaus Berlin (Other); Universität des Saarlandes (Other); University of Padova (Other); Masaryk University (Other); University of Budapest (Other); Hospital Universitari de Bellvitge (Other); Hospital General Universitario Gregorio Marañon (Other); Neurosurgical Department, Clinique St. Jaen, Brussels, Belgium (Unknown)
Responsible Party: Prof. Dr. med. Petra M. Klinge, International Neuroscience Institute Hannover
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: european-nph-study-01; Dr.Klinge.C.T.Agreement08/2004; Dr.Klinge.C.T.Agreement10/2006
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: normal pressure hydrocephalus; cerebrospinal fluid dynamic test; cerebrospinal fluid outflow resistance; cerebrospinal compliance; outcome; shunt surgery; normal pressure hydrocephalus guidelines; biomarkers; shunt surgery selection; Outcome measures; Outcomes assessment; Outcome and process assessment
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Ventriculoperitoneal Shunt

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ventriculo-peritoneal Shunt — Surgical implantation of a ventriculo-peritoneal cerebrospinal fluid shunt with an adjustable valve system using the Codman-Hakim programmable valve system [pressure settings: 30 - 200 mmH20]
  Other Names: see above

SUMMARY:
The purpose of the study is to determine the predictive values and prognostic accuracies of CSF dynamic measures, the TAP -TEST (high-volume cerebrospinal fluid withdrawal), resistance to CSF outflow and compliance in the prediction of shunt-treatment outcome in patients with idiopathic normal pressure hydrocephalus.

DETAILED DESCRIPTION:
Study background:

The selection of patients with idiopathic normal pressure hydrocephalus (INPH) for shunting remains difficult. The upcoming guidelines for the diagnosis and management of INPH state that there is no accepted standard for the clinical presentation, the results of imaging and the various tests that provide information on CSF dynamics 1. Hebb and Cusiamo could not find a single test that reliably predicts outcome after shunting in their systematic review of INPH 2. To properly evaluate the predictive value of diagnostic tests for the outcome of shunting all patients should receive a shunt irrespective of the test results. Only a few studies set up to examine the diagnostic reliability of tests of CSF dynamics fulfilled this condition. The common finding of these studies was that the predictive value of a positive test was high but the negative predictive values were disappointingly low.

In the Dutch Normal Pressure Hydrocephalus Study, containing 101 patients, the positive and negative predictive values of lumbar constant flow infusion were 92% and 34% for an Rout of 18 mmHg/ml/min and 100% and 27% for an Rout of 24 3. External lumbar CSF drainage for 4 days resulted in positive and negative predictive values of 87% and 36% 4. The predictive value of the cerebrospinal fluid tap test reported by Wikkelso et al in 1986 was 100% for a positive and 45% for a negative test 5 Another parameter of CSF dynamics is elastance that can be expressed by the pressure volume-index (PVI). In a group of 30 patients with NPH high elastance, i.e low PVI was the best predictor of a marked and rapid reduction of ventricular size after shunting 6.

One of the major issues is whether the false negative tests mostly occur in the same population. In these patients the INPH might be caused not so much by a CSF circulation disorder but by parenchymal disease. From our clinical experience we think that different patients have false negative tests, we frequently encounter cases with a positive tap test and a negative infusion test or the reverse. This is also shown in a study by Kahlon et al. who performed an infusion test and a tap test in 68 patients suspected of NPH. Both tests agreed in only 45% and they were both negative in 31% of patients 7.

An important drawback of all INPH studies so far is the rather limited number of patients and, the "mixing" of idiopathic NPH patients (primary NPH) with those of known cause (secondary NPH) such as trauma, subarachnoid hemorrhage and stroke.INPH is considered a multfactorial condition with a disturbance of CSF circulation as well as parenchymal abnormalities in a vulnerable population with much comorbidity. Because of the many outcome variables a study on the prediction of outcome needs large numbers of INPH patients. With a few exceptions, previous studies on CSF dynamics in INPH were conducted in single high quality institutions. We also have to demonstrate that the same or even better results can be obtained with international cooperation providing higher patients numbers. Therefore we intend to conduct a large European multicentre study on INPH including at least 200 patients. All these patients will receive the same shunt system and will be followed-up by a standardized protocol using primary and secondary NPH outcome measures. Because of the continuing controversy with respect to the appropriate shunt opening pressure and the many problems of over- and underdrainage after insertion of the shunt, we chose the Codman Hakim programmable valve 8.

STUDY AIMS

To determine primarily the sensitivity, specificity, positive- and negative predictive value of resistance to outflow of CSF (Rout) and the CSF-Tap-Test for prediction of the effect of shunt surgery in patients with idiopathic NPH (INPH) by a prospective "blinded" confirmative study.

Secondarily the predictive value of elastance and CSF biochemical markers will be evaluated in the same population.

Further, the predictive value of other tests as rCBF and vascular reserve capacity (PET or SPECT), MR investigations (i.e. fMRI, MRS and/or diffusion tensor imaging etc.), continuous CSF drainage, B-wave analyses and other investigations can be evaluated by cooperation between individual centres.

General study design:

A prospective "blinded" confirmative study of at least 200 consecutively included patients with INPH fulfilling the clinical and radiological inclusion and exclusion criteria. Patients will be included during a period of 2 years by 20 or more centres that will enrol at least 5 patients per year each. All patients in the study will receive a ventriculo-peritoneal shunt, using the Codman Programmable valve.

After inclusion but prior to surgery 4 obligatory tests will be performed. We will measure the resistance to outflow of CSF (Rout) and the intracranial elastance, a CSF-Tap-Test will be carried out and CSF biochemical markers are determined. The caretakers are blinded for these results. Rout and the results of the tap test are the primary investigations.

Optional tests as rCBF and vascular reserve capacity (PET or SPECT), MR investigations (i.e. fMRI, MRS and/or diffusion tensor imaging ), continuous CSF drainage and B-wave analyses will also be performed prior to surgery. The number of patients included in a study of an optional test should be at least 30 in order to qualify for recording of the data in the database.

The patients are evaluated by a battery consisting of a handicap scale (modified Rankin scale) and 7 tests that measure gait, cognition and bladder function, before and 3 and 12 months after surgery or establishment of a working shunt. The patients are also checked one month after surgery to secure shunt efficacy.

The changes in clinical signs and disability after surgery are correlated to the results of the obligatory and optional tests. The primary outcome measures are the differences between the pre-operative and 12 months scores in the Rankin Scale and the composite NPH scale. These will be correlated with the results of the two primary investigations, resistance to CSF outflow (mmHg/ml/min) and CSF Tap Test (% change).

Patients data will be stored electronically in a web-based central data base using a special data security system for data transfer. Access to the database will be provided through an official homepage protected by a certified username/password based authenticity mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis (neurological and radiological criteria) of idiopathic normal pressure hydrocephalus

Typical INPH

Clinical criteria:

* Gradually developed gait disturbance of both legs, unexplained by other conditions. Disturbance of tandem walking, multi-step turning, small steps and wide base must be present at least.
* MMSE score 21-30 without aphasia, apraxia and agnosia
* Bladder instability and postural instability may be present.

Radiological criteria (MRI):

* Symmetrical communicating quadri-ventricular enlargement without cortical infarcts or other clinically relevant parenchymal lesions but lacunar infarcts of less than 1 cc may be present
* Evans index > 0.30 and temporal horns and third ventricle relatively enlarged.
* Mild cortical atrophy and mild leuco-araiosis may be present.

Questionable NPH

Clinical criteria:

* Any gait disturbance of both legs that does not fulfill the criteria of typical INPH, but is compatible with INPH.
* MMSE score < 21
* Bladder instability and postural instability may be present.

Radiological criteria (MRI):

* Symmetrical communicating quadri-ventricular enlargement without major parenchymal lesions. Single cortical infarcts and lacunar infarcts may be present.
* Evans index > 0.30.
* Moderate cortical atrophy and moderate to severe leuco-araiosis may be present.

Exclusion Criteria:

* Secondary Normal pressure Hydrocephalus
* Non-communicating hydrocephalus
* Secondary NPH (after SAH, trauma, infection, neurosurgical procedure). Trauma or infection are regarded as relevant if the patient was unconscious in relation to the trauma or required hospitalisation for his meningo-encephalitis.
* INPH-patients later shown to have ICP > 18 mm Hg.
* Contra-indications to surgery.
* Patients refusing shunt surgery
* Restricted life-expectancy
* Patients not capable of managing the tests or investigations at entry of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2004-10; Primary Completion 2008-03 (Actual); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 12 months

SECONDARY OUTCOMES:
Neuropsychological measures (Stroop test, REy-auditory verbal learing test, PEG-BOARD TEST), Balance -score, Incontinence-score, Gait-score, Walking-score | three and 12 months
Balance -score | three and 12 months
Incontinence-score | three and 12 months
Gait-score | three and 12 months
Walking-score | three and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Petra M Klinge, MD, Principal Investigator — International Neuroscience Institute Hannover; Carsten I Wikkelsoe, MD, Principal Investigator — Sahlgrenska University, Gothenburg, Sweden; Jos TH Tans, MD, Principal Investigator — Westeinde Hospital, Den Haag, Netherlands
Locations (1):
- International Neuroscience Institute Hannover, Hanover, Lower Saxony, Germany

REFERENCES:
- [Background] Marmarou A, Black P, Bergsneider M, Klinge P, Relkin N; International NPH Consultant Group. Guidelines for management of idiopathic normal pressure hydrocephalus: progress to date. Acta Neurochir Suppl. 2005;95:237-40. doi: 10.1007/3-211-32318-x_48. PMID 16463856
- [Background] Hebb AO, Cusimano MD. Idiopathic normal pressure hydrocephalus: a systematic review of diagnosis and outcome. Neurosurgery. 2001 Nov;49(5):1166-84; discussion 1184-6. doi: 10.1097/00006123-200111000-00028. PMID 11846911
- [Background] Boon AJ, Tans JT, Delwel EJ, Egeler-Peerdeman SM, Hanlo PW, Wurzer HA, Avezaat CJ, de Jong DA, Gooskens RH, Hermans J. Dutch normal-pressure hydrocephalus study: prediction of outcome after shunting by resistance to outflow of cerebrospinal fluid. J Neurosurg. 1997 Nov;87(5):687-93. doi: 10.3171/jns.1997.87.5.0687. PMID 9347976
- [Background] Walchenbach R, Geiger E, Thomeer RT, Vanneste JA. The value of temporary external lumbar CSF drainage in predicting the outcome of shunting on normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2002 Apr;72(4):503-6. doi: 10.1136/jnnp.72.4.503. PMID 11909911
- [Background] Wikkelso C, Andersson H, Blomstrand C, Lindqvist G, Svendsen P. Normal pressure hydrocephalus. Predictive value of the cerebrospinal fluid tap-test. Acta Neurol Scand. 1986 Jun;73(6):566-73. doi: 10.1111/j.1600-0404.1986.tb04601.x. PMID 3751498
- [Background] Tans JT, Poortvliet DC. Reduction of ventricular size after shunting for normal pressure hydrocephalus related to CSF dynamics before shunting. J Neurol Neurosurg Psychiatry. 1988 Apr;51(4):521-5. doi: 10.1136/jnnp.51.4.521. PMID 3379425
- [Background] Kahlon B, Sundbarg G, Rehncrona S. Comparison between the lumbar infusion and CSF tap tests to predict outcome after shunt surgery in suspected normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2002 Dec;73(6):721-6. doi: 10.1136/jnnp.73.6.721. PMID 12438477
- [Background] Zemack G, Romner B. Adjustable valves in normal-pressure hydrocephalus: a retrospective study of 218 patients. Neurosurgery. 2002 Dec;51(6):1392-400; discussion 1400-2. PMID 12445344
- [Derived] Wikkelso C, Hellstrom P, Klinge PM, Tans JT; European iNPH Multicentre Study Group. The European iNPH Multicentre Study on the predictive values of resistance to CSF outflow and the CSF Tap Test in patients with idiopathic normal pressure hydrocephalus. J Neurol Neurosurg Psychiatry. 2013 May;84(5):562-8. doi: 10.1136/jnnp-2012-303314. Epub 2012 Dec 18. PMID 23250963